CLINICAL TRIAL: NCT05747690
Title: A Randomized, Controlled, Split-Face Study to Evaluate the Clinical Performance and Safety of Intradermal Injection of KIO015 for Tissue Filling in Subjects With Signs of Cutaneous Dehydration on the Face
Brief Title: Evaluation of Performance and Safety of KIO015 in Face Tissue Filling
Acronym: PLUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kiomed Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20E1676-2/PLUM
Record Dates: First submitted 2023-01-16; First posted 2023-02-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Skin Quality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KIO015 - Cohort 1 (Experimental): One injection of KIO015 on the hemi-face. The untreated hemi-face is used as a comparator.
  Interventions: Device: KIO015
- KIO015 - Cohort 2 (Experimental): 3 injections at one month interval on the hemi-face. The untreated hemi-face is used as a comparator.
  Interventions: Device: KIO015

INTERVENTIONS:
Device: KIO015 — Innovative carboxymethyl chitosan-based biomaterial intended for intradermal injection

SUMMARY:
The clinical investigation is designed to primarily confirm the performance of KIO015 in improving the GAIS assessment, a subjective parameter, including skin roughness. A non-treated zone (untreated hemi-face) was used as comparator for exact evaluation of the zones between the treated and untreated ones The safety of KIO015 was also evaluated for confirmation of initial data.

For this purpose, 78 healthy subjects were injected in half of the face. In KIO015-PLUM, healthy subjects with signs of cutaneous aging and dehydrated skin on the face received either one or three dermal injections:

* Cohort 1: one intradermal injection session of KIO015 device on M0, to evaluate the effect of a single injection session
* Cohort 2: three intradermal injection sessions of KIO015 device on M0, M1 and M2, to evaluate the effect of 3 injection sessions as performed for state-of-the-art products.

ELIGIBILITY:
Inclusion Criteria:

* Subject with signs of cutaneous ageing on the face according to investigator's judgment.
* Subject with dehydrated skin on the face (value < 60 A.U with Corneometer®).
* Subject having given freely and expressly his informed consent.
* Subject, psychologically able to understand the study related information and to give a written informed consent.
* Subject affiliated to a health social security system.
* Female of childbearing potential must use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study and during all the study.
* Female subjects of childbearing potential must have a negative pregnancy test at the inclusion.

Exclusion Criteria:

In terms of population

* Pregnant or nursing woman or planning a pregnancy during the study.
* Woman with menopause from less than 1 year or in perimenopause, without hormonal treatment.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* Subject participating to another research on human beings or being in an exclusion period for a previous study.
* Subject having received 4500 euros indemnities for participation in research involving human beings in the 12 previous months, including participation in the present study.
* Subject suffering from dysmorphophobia or having an unreasonable expectation about the treatment results.
* Intensive exposure to sunlight or UV-rays within the previous month and foreseen during the study.
* Subject with a tattoo, a scar, moles or too many hairs or anything on the face which may interfere with the study at the investigator appreciation.
* Subject having resorbable filling product (e.g., hyaluronic acid) injections, a laser treatment, an ultrasound-based treatment a dermabrasion, a surgery, a deep chemical peeling or other ablative procedure on the face within the past 12 months prior to study start.
* Subjects having received botulinum toxin in the face within the 6 previous months.
* Subject having received mesotherapy products in the face within the 3 previous months.
* Subject having done a superficial or medium peeling or a superficial scrub on the face within the 2 previous months.
* Subject using cosmetic products with alpha hydroxy acids (AHA).
* Subject with subcutaneous retaining structure on the face (meshing, threads, gold strand).
* Subject having received injections of permanent (e.g., acrylate polymers, silicone, polytetrafluoroethylene) or semi-permanent filling on the face.
* Subject with an excessive consumption of alcohol (more than 2 glasses of wine per day) and/or tobacco (more than 10 cigarettes per day).

In terms of associated pathology

* Subject with ongoing and/or uncontrolled and/or recently recovered (<6 months) depression or psychiatric disorders or any other disorder that may pose a health risk to the subject in the study and/or may have an impact on the study assessments.
* Subject with severe, ongoing and uncontrolled diseases such as malignancy or history of malignancy, type I diabetes, liver failure, renal failure, lung/heart disease, neoplasia, malignant blood disease, tumor, HIV, or other major disease (e.g., systemic fungal infection).
* Subject with recurrent porphyria, coronary insufficiency, ventricular rhythm disorders, severe hypertension, obstructive cardiomyopathy, hyperthyroidism.
* Subject with any skin or systemic disease (acute and/or chronic), in the previous year, likely to interfere with the measured parameters or to put the subject to an undue risk.
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
* Subject with current cutaneous inflammatory or infectious processes (e.g., acne, herpes, mycosis, papilloma, chronic eczema, atopic dermatitis …), abscess, unhealed wound, or a cancerous or precancerous lesion on the face.
* Subject with multiple allergies, anaphylactic shock history, evolutive allergic pathologies.
* Subject having history of allergy or hypersensitivity to one of the components of the tested device
* Subject having history of hypersensitivity to lidocaine and/or prilocaine or local anaesthetics of amide type or one of the excipients of EMLA® 5% cream.
* Subject having history of hypersensitivity to chlorhexidine (or similar product) or one of the excipients of alcoholic chlorhexidine 0.5%.
* Subject predisposed to keloids or hypertrophic scarring.
* Subject with coagulation and/or homeostasis disorders.
* Subject with pigmentation disorders. Related to previous or ongoing treatment
* Subject under anti-coagulant treatment (such as aspirin, nonsteroidal anti-inflammatory drugs) or treatment liable to interfere with the healing process or hemostasis, during the previous month and during the study
* Subject receiving any treatment that, in the opinion of the clinical investigator, may interfere with test results or put the subject to undue risk.
* Subject undergoing a topical (on the face) or systemic treatment:

  * anti-inflammatory medication and/or anti-histamines during the previous 2 weeks and during the study;
  * immunosuppressors and/or corticoids during the 4 previous weeks and during the study;
  * retinoids during the 6 previous months and during the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Global aesthetic improvement with GAIS (Global Aesthetic Improvement Scale) | 1 month after the first intradermal injection for both cohorts.
  Clinical evaluation of global aesthetic improvement of the treated area with GAIS (Global Aesthetic Improvement Scale) evaluated by the investigator. Comparison to a non-treated zone.

SECONDARY OUTCOMES:
For both cohorts combined, evaluation of cutaneous hydration in a sub-group of subjects not using hydrating agent | 1 month after the first intradermal injection
Change from baseline of epidermis hydration with Corneometer® | 1 month, 2 months, 3 months, 6 months, 9 months and 12 months (cohort 1 only) after each injection session.
  For each cohort, change from baseline of epidermis hydration of the treated zone measured with Corneometer®
Change from baseline of dermis hydration with Moisturemeter D® | 1 month, 2 months, 3 months, 6 months, 9 months and 12 months (cohort 1 only) after each injection session.
  For each cohort, change from baseline of dermis hydration of the treated zone measured with Moisturemeter D®
Change from baseline of skin oxidative stress | 7 days (cohort 1 only), 1 month, 3 months and 6 months after each injection session.
  For each cohort, change from baseline of skin oxidative stress from skin superficial sampling on the treated area at the different time points and comparison to a non-treated zone.
Change from baseline of epidermis hydration compared to a non-treated zone with Corneometer® | At 1 month, 2 months, 3 months, 6 months and 9 months after the last injection session in both cohorts
  Comparison of both cohorts for the change from baseline compared to a non-treated zone of Corneometer®
Change from baseline of dermis hydration compared to a non-treated zone with Moisturemeter® | At 1 month, 2 months, 3 months, 6 months and 9 months after the last injection session in both cohorts
  Comparison of both cohorts for the change from baseline compared to a non-treated zone of Moisturemeter®
Change from baseline of skin oxidative stress compared to a non-treated zone | At 1 month, 2 months, 3 months and 6 months after the last injection session in both cohorts
  Comparison of both cohorts for Change from baseline of skin oxidative stress compared to a non-treated zone
For both cohorts combined, change from baseline of epidermis hydration of the treated zone, measured with Corneometer® and comparison to a non-treated zone | 1 month after the first injection
For both cohorts combined, change from baseline of dermis hydration of the treated zone, measured with Moisturemeter D® and comparison to a non-treated zone | 1 month after the first injection
Global aesthetic improvement with GAIS (Global Aesthetic Improvement Scale) | 7 days, 1 month, 2 months, 3 months, 6 months, 9 months and 12 months (cohort 1 only) after each injection session.
  Clinical evaluation of global aesthetic improvement of the treated area with GAIS (Global Aesthetic Improvement Scale) evaluated by the investigator. Comparison to a non-treated zone.
Pain felt by the subject using a subjective evaluation questionnaire | Immediately after the injection session.
  Evaluation of pain felt by the subject using a subjective evaluation questionnaire on skin improvement of the treated area.
Subject satisfaction using a subjective evaluation questionnaire | 1 month, 2 months, 3 months, 6 months, 9 months and 12 months (cohort 1 only)
  Evaluation of subject satisfaction using a subjective evaluation questionnaire on skin improvement of the treated area.
Difference in Global aesthetic improvement with GAIS (Global Aesthetic Improvement Scale) between Cohorts 1 and 2 | At 1 month, 2 months, 3 months and 6 months after the last injection session in both cohorts
  Comparison of percentage of subjects with an improvement of the GAIS (Global Aesthetic Improvement Scale) of the treated area, evaluated by the investigator between cohort 1 and 2
Difference in subject satisfaction between Cohorts 1 and 2. | At 1 month, 2 months, 3 months and 6 months after the last injection session in both cohorts
  Comparison of percentage of satisfied subjects using a subjective evaluation questionnaire on skin improvement of the treated area between cohort 1 and 2
Appreciation of the injection quality using a subjective evaluation questionnaire | Immediately after the injection sessions
  Evaluation of the appreciation of the injection quality using a subjective evaluation questionnaire completed by the injectors
Evaluation of injection site reactions (investigator) | 7 days, 1 month, 2 months, 3 months, 6 months, 9 months and 12 months (cohort 1 only)
  Percentage of injection site reactions recorded by the investigator
Evaluation of injection site reactions (subject) | During 30 days after each injection session.
  Evaluation of the duration and severity of the injection site reactions by the subject recorded in a diary.
Product safety | Through study completion, up to 12 months
  Collection of adverse events and concomitant treatments

OTHER OUTCOMES:
Needle size | 1 month, 2 months, 3 months, 6 months and 9 months
  Comparison of the two sub-groups using different needles (30G and 32G)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia MOREL-MANDRINO, MD, Principal Investigator — Eurofins Dermscan Pharmascan
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No